CLINICAL TRIAL: NCT02372708
Title: Clinical Research on the Treatments on Advanced Malignant Melanoma by Combining in Situ Immunotherapy and Laser Therapy
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, DuNan, professor, Chinese PLA General Hospital
Other Study IDs: ML125396
Record Dates: First submitted 2015-02-13; First posted 2015-02-26 (Estimated); Last update posted 2015-02-26 (Estimated); Status verified 2015-02

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Radiation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Experimental: diluted dinitrophenyl(DNP) Vaseline (which equaled to 2% DNP 0.1ml) was started to be directly spread on the surfaces of primary or metastatic tumors of malignant melanoma patients since the first day of every circle of chemotherapy, simultaneously laser irradiation was carried out for 10 min, the power density of laser irradiation was 1W/cm2. The tumors were wrapped and blocked for two days to induce contact dermatitis. If lymph nodes had been cleared, sensibilization of 2×2cm was performed at occipital region. It was repeated once a week.
  Interventions: Drug: dinitrophenyl(DNP); Radiation: Radiation
- Control: only diluted DNP Vaseline was spread and the operation were the same with the treatment group
  Interventions: Drug: dinitrophenyl(DNP)

INTERVENTIONS:
Drug: dinitrophenyl(DNP)
Radiation: Radiation — laser irradiation was carried out for 10 min, the power density of laser irradiation was 1W/cm2
  Groups: Experimental

SUMMARY:
To evaluate the therapeutic efficacy and the safety for the treatments on malignant melanoma by combining semiantigen dinitrophenyl (DNP) in situ immunotherapy and laser therapy, and carry out monitoring on related immunological parameters of the patients.

72 patients with stage III (b or c) or stage IV skin (which could not be excised by operations) malignant melanoma were treated by combining simple semiantigen DNP in situ immunotherapy and laser therapy respectively. The changes in peripheral blood CD4+CD25+Treg regulatory T cells (Treg), CD8+T, CD4+ T effector cells, IL-10, TGF-β and other inhibitory cytokines of the patients were detected, the changes in anti-DNP IgG antibody titer was monitored, the relationship between delayed-type hypersensitivity (DTH) and survival was observed, and results of clinical follow-ups were also examined.

ELIGIBILITY:
Inclusion Criteria:

* pathologically diagnosed as malignant melanoma, HMB45 (+～++++), S100 (+～++++);
* Basically normal hepatic and renal functions as well as results for blood routine examinations;
* Karnofsky score ≥ 60;
* Anticipated life span for more than three months;
* They were all malignant melanoma patients suffering from skin malignant melanoma of local or distal metastasis unsuitable for operations in their skin;
* The therapeutic efficacy was objectively evaluated with reference to the criteria from WHO;
* All of the subjects had signed the informed consent and had been submitted and approved by the ethic committee of the hospital, the compliance was good and follow-ups can be easily carried out.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with stage III (b or c) or stage IV skin (which could not be excised by operations) malignant melanoma
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2008-08; Primary Completion 2012-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
ORR | 6 weeks after administration whose achieve CR and PR
  Patients who have complete regression or partial regression

SECONDARY OUTCOMES:
PFS | From enrollment to progression or death, which up to 2 years
OS | From enrollment to death, which up to 2 years
biomarker (peripheral blood CD4+CD25+Treg regulatory T cells (Treg), CD8+T, CD4+ T effector cells, IL-10, TGF-β) | day 0 and day 2,5,10,20
  peripheral blood CD4+CD25+Treg regulatory T cells (Treg), CD8+T, CD4+ T effector cells, IL-10, TGF-β

CONTACTS AND LOCATIONS:
Overall Officials: Nan Du, PHD, Principal Investigator — First Affiliated Hospital, Chinese PLA General Hospital
Locations (1):
- First Affiliated Hospital, Chinese PLA General Hospital, Beijing, Beijing Municipality, China